CLINICAL TRIAL: NCT04042168
Title: Implications of Appropriate Use of Inhalers in Chronic Obstructive Pulmonary Disease (COPD)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No subject met criteria for enrollment and study was stopped due to the pandemic
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Surya P Bhatt, Associate Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300003947
Record Dates: First submitted 2019-05-30; First posted 2019-08-01 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Inhalers
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: UAB Pulmonary Clinic Patients with history of COPD
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Inappropriate use of inhalers and medication change. Pre-post intervention data will be compared.
  Interventions: Diagnostic Test: In Check Dial test

INTERVENTIONS:
Diagnostic Test: In Check Dial test — In Check Dial test will test the ability to actuate the inhaler.

SUMMARY:
Using various types of inhalers is the treatment cornerstone for COPD patients to control their symptoms. Many inhaler devices require minimum inspiratory effort to activate the device, COPD patients commonly use such devices. Those devices deliver the medications only when the patient forcefully inhales so the drug can reach the lungs, thus exerting their therapeutic action. The effect of appropriate use of the inhalers in patients with COPD is not well studied, and the impact of demonstrating that a patient can inhale forcefully enough to activate a device on its' effect on symptoms is also lacking in the medical literature. The purpose of this study is to find out:

1. the frequency of COPD patients demonstrating an appropriate use of inhalers that have flow-triggered systems,
2. whether the appropriate use of inhalers impacts the Quality of Life and Shortness of Breath of COPD patients, and
3. the impact of appropriate use of inhalers on FEV1 in COPD patients.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a chronic systemic inflammatory disease associated with substantial morbidity and mortality and is now the 3rd leading cause of death in the United States. The majority of COPD-related symptoms are managed using inhaled therapy. Inhalation is a safe, efficacious and quick way for drug delivery. Inhaled therapy permits direct availability of the active drug to the lungs, requiring lower doses of the drug and causing lower systemic side effects as compared to oral therapy. There are four major types of inhalation devices: pressurized metered-dose inhalers (MDI), dry powder inhalers (DPI), soft mist inhalers (SMI), and nebulizers. Every type has its advantages and disadvantages that are important to understand to determine their suitability for COPD patients. Despite that, choosing the appropriate device for patients remains a challenge for the prescribing physician.

For all inhaler devices, training patients on how to use them appropriately is required to attain ideal therapeutic benefits. Multiple studies have estimated that about 28-68% of patients were inappropriately using their inhalation devices to benefit from the prescribed drug. Brocklebank et al. performed a systematic review looking at the effectiveness of inhaler device use in COPD and asthma patients. They found that ideal inhaler scores were reached by 59% of subjects with DPIs and 43% with MDIs. 5 on the other hand, the aggregate data from this systematic review showed that after teaching the correct technique there was no difference in patients' ability to use DPI or MDIs. One of the common problems leading to inappropriate use of the inhalation devices is breath asynchrony. An in-vitro study done by Wilkes et al. showed that breath asynchrony significantly decreases the mass of medication inhaled from an MDI. It showed that actuation of only one second earlier to inhalation decreases the inhaled mass of medication by about 90%. Likewise, actuation later on in the inspiratory cycle could lead to filling the anatomic dead space with the aerosolized medication. This issue seems to be less pronounced in DPI devices, as those systems are mainly passive in their function depending on the mechanical effort of the patient to release the medication and supply it to the effective areas inside the lungs through inspiration. On the other hand, there seem to be multiple factors leading to suboptimal use of DPIs such as the inability to activate the device with enough inspiratory effort.

Very limited studies looked at the inspiratory effort for COPD patients and the efficacy of inhaler use. Burnell et al. looked at the performance of 17 COPD patients with severe obstruction using an inhalation simulator to establish dosing performance of the Diskus inhaler with fluticasone and Turbuhaler inhaler with budesonide. Peak inspiratory flow was significantly higher through the Diskus as compared with Turbuhaler (mean 82.3 l/min vs 53.5 l/min, P < 0.001). Also, the Diskus inhaler was shown that drug delivery was more dependent on peak inspiratory flow with the Turbuhaler than with the Diskus. On the other hand, a study looked at the performance of a high resistance inhaler (HandiHaler) in 26 men with stable COPD. Patients were categorized into 3 groups of severity, based on their predicted FEV-1(less than 27%, 28 - 45%, and more than 46%) and then measured the inspiratory flow through the HandiHaler. The median peak inspiratory flow rates for each group were 45, 45.6, and 35.4 L/min respectively. The minimum peak inspiratory flow rates were 28.2, 21.6 and 20.4 L/min. The authors then conducted an in-vitro analysis to assess the minimum inspiratory flow rate indicated for the delivery of the medication and found to be at flow rates as low as 20 l/min. They concluded that drug delivery was adequate despite the severity of COPD. Up to our knowledge, no previous studies looked at the change of symptoms control in-vivo in relation to the inhalation effort of COPD patients and the appropriate use of their inhalers.

The investigators hypothesize that COPD patients with high peak inspiratory flow rates and appropriate use of inhalers device have better symptoms control with using breath-actuated inhalers as compared to patients who fail to actuate inhalers devices (inappropriate use of inhalers) and have low peak inspiratory flow.

The investigators have designed a prospective study to determine the inspiratory effort status and the change of symptoms in stable COPD patients seen as outpatient. Pulmonary function testing, COPD related quality of life and shortness of breath will be assessed at baseline and 3 months after obtaining the status of inhalers use at baseline.

ELIGIBILITY:
Inclusion Criteria:

* provide informed consent
* age 40 and older
* history of COPD
* screen at pulmonology clinic
* on at least one maintenance inhaler

Exclusion Criteria:

* Patients with a secondary diagnosis of congestive heart failure and other respiratory conditions that the investigators deem could confound the diagnosis including but not limited to pneumonia
* bronchiectasis and lung cancer will be excluded
* pregnant or breastfeeding women will be excluded
* patients with conditions that preclude an adequate peak inspiratory flowmetry including but limited to facial deformities
* neurologic disorders precluding command following
* trachestomy dependent patients

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2022-08-09 (Actual); Study Completion 2022-08-09 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with COPD on inappropriate inhalers | Baseline
  The frequency of COPD patients demonstrating an inappropriate use of inhalers that have flow-triggered systems
Change in St George's Respiratory Questionnaire (SGRQ) Score in 3 months | 3 months
  Whether the appropriate use of inhalers impacts the quality of life and symptom control of COPD patients. SGRQ score ranges from 0 to 100, higher the score worse the quality of life. A change of 4 units is considered the minimum clinically important difference.
Change in the forced expiratory volume in the first second (FEV1) in 3 months | 3 months
  Whether the appropriate use of inhalers impacts the lung function of COPD patients.
Change in shortness of breath in 3 months measured using the San Diego Shortness of breath Questionnaire. | 3 months
  Whether the appropriate use of inhalers impacts shortness of breath in COPD patients. The Shortness of Breath Questionnaire score ranges from 0 to 100, higher the score worse the quality of life. A change of 5 units is considered the minimum clinically important difference.

CONTACTS AND LOCATIONS:
Locations (1):
- UAB Department of Medicine, Pulmonary Division, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No